CLINICAL TRIAL: NCT05218746
Title: Comparison Between Serratus Anterior Plane Block Versus Erector Spinae Plane Block for Postoperative Analgesia After Video-Assisted Thoracoscopic Surgery
Brief Title: Regional Blocks for Postoperative Analgesia After Video-Assisted Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Beshoy Aziz, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Regional blocks in VATS
Record Dates: First submitted 2022-01-31; First posted 2022-02-01 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus anterior block (Experimental): Regional analgesic block of anterolateral chest wall
  Interventions: Procedure: Serratus anterior plane block
- Erector spinae block (Experimental): Regional analgesic block for the whole chest wall
  Interventions: Procedure: Erector spinae block

INTERVENTIONS:
Procedure: Serratus anterior plane block — High-frequency linear transducer will be placed on the patient's midaxillary line in the transverse plane, at the level of the fifth rib, with the indicator oriented toward the operator's left. With the rib, pleural line, and overlying serratus anterior and latissimus dorsi muscles visualized, Then, using ultrasound guidance, the needle will be advanced in-plane at an angle of approximately 45 degrees towards the fifth rib . one millileter normal saline will be injected to confirm placement and to hydro-dissect the fascial layers and open the potential space.
  Arms: Serratus anterior block
Procedure: Erector spinae block — A high-frequency linear ultrasound probe will be placed in a longitudinal orientation 3 cm from the midline. Once the erector spinae muscle and the transverse processes is identified, spinal needle will be inserted in a caudad-to-cephalad direction until the tip lay in the interfacial plane deep to the erector spinae muscle.
  Arms: Erector spinae block

SUMMARY:
The aim of this study is to compare serratus anterior plane block and erector spinae plane block for postoperative analgesia after VATS as measured by the duration till 1st requirement of analgesia.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery has become the standard surgical procedure for both minor and major oncological lung surgery, as it is considered less invasive and equally effective compared with thoracotomy . However, it is a fact that pain following VATS can be severe and long-lasting. According to Homma et al., 18.8% of patients who undergo VATS present with persistent pain 2 months after surgery.

Serratus anterior plane block is a type of interfascial plane block that was defined by Blanco and his colleagues in 2013 .Ultrasound-guided SAPB has recently gained the interest of the anesthesiologists and pain physicians due to its efficacy, relative ease, single-injection method with limited side-effect profile.

The SAPB targets the lateral cutaneous branches of the thoracic intercostal nerves, which arise from the anterior rami of the thoracic spinal nerves and run in a neurovascular bundle immediately inferior to each rib. At the midaxillary line, the lateral cutaneous branches of the thoracic intercostal nerve traverse through the internal intercostal, external intercostal, and serratus anterior muscles innervating the musculature of the lateral thorax.These branches of the intercostal nerves, therefore, travel through the two potential spaces described above. Local anesthetic inserted into these planes will spread throughout the lateral chest wall, resulting in paresthesia of the T2 through T9 dermatomes of the anterolateral thorax.

Erector spinae plane block is an interfascial plane block that was defined by Forero and colleagues in 2016. Erector spinae plane block has a wide indication range for pain management of the thoracic, abdominal , lumbar, hip, and even shoulder areas . Erector spinae plane block is a paraspinal block that targets the dorsal and ventral rami so that it can provide analgesia in the anterolateral and posterior chest wall .

Erector spinae plane block emerged in recent years to be effective in reducing postoperative pain at 24 h, i.e. preoperative ESPB plus intravenous opioid reduced pain scores and opioid consumption after VATS when compared with intravenous fentanyl only .

ELIGIBILITY:
Inclusion criteria

* Patients with American Society of Anesthesiologists (ASA) physical status 1-3 --
* scheduled for VATS .

Exclusion Criteria:

1. ≤20 or ≥80 years old.
2. Refusing to participate in the study .
3. History of allergy to the medications used in the study.
4. Contraindication to regional anesthesia (including coagulopathy and local infection).
5. Severe hepatic impairement (serum protein < 3g/dl and serum bilirubin > 3mg/dl) .
6. Renal dysfunction (as determined by creatinine levels greater than 2mg/dl or predicted creatinine clearance (CLcr)<50ml/min).
7. Psychiatric disorder.
8. Pregnancy.
9. Body mass index (BMI) ≥40 or ≤18 kg/m2.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
the duration till 1st requirement of analgesia | postoperative first day
  The time from the end of the operation till Visual analogue score more than 3

SECONDARY OUTCOMES:
Analgesic consumption | postoperative first day
  Total analgesic opioid consumption during the first postoperative day

IPD SHARING:
Plan to Share IPD: No